CLINICAL TRIAL: NCT00181610
Title: Recombinant Human Prolactin for Lactation Induction in Mothers of Premature Infants
Brief Title: Recombinant Human Prolactin for Lactation Induction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Corrine Welt, Associate Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2001P001475
Record Dates: First submitted 2005-09-09; First posted 2005-09-16 (Estimated); Results first posted 2013-05-10 (Estimated); Last update posted 2018-01-03 (Actual); Status verified 2017-12

CONDITIONS: Lactation
Keywords: Lactation; Breastfeeding; Premature infants; Prolactin; Primary lactation insufficiency
MeSH Terms: conditions — Breast Feeding; Premature Birth | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Placebo group normal saline twice per day
  Interventions: Biological: Normal Saline
- 2 (Active Comparator): Recombinant human prolactin 60 mcg/kg every 12 hours
  Interventions: Drug: Recombinant Human Prolactin
- 3 (Active Comparator): Recombinant human prolactin 60 mcg/kg alternating with normal saline placebo every 12 hours
  Interventions: Biological: Recombinant human prolactin; Biological: Normal Saline

INTERVENTIONS:
Drug: Recombinant Human Prolactin — 60 mcg/kg every 12 hours
  Arms: 2
Biological: Recombinant human prolactin — 60 mcg/kg given every 12 hours or every 24 hours
  Arms: 3
Biological: Normal Saline — twice per day
  Arms: 1; 3

SUMMARY:
The purpose of the study is to assess the safety and determine the effects of the hormone prolactin on lactation (breast milk production).

DETAILED DESCRIPTION:
The study is a randomized, double blind, placebo controlled trial. Subjects will be admitted to the General Clinical Research Center (GCRC) as outpatients to undergo their baseline pumping study. One lactation consultant will educate all subjects in the proper technique for pumping on the first day of the study and will evaluate their technique on day 5 and day 8 of the study. The lactation consultant will also instruct patients to record the volume of milk pumped and the time of each pumping episode. Subjects will be encouraged to have direct contact with their infants prior to pumping. All infant contact, infant latching onto the breast and mother's stress level will also be recorded throughout the study. Starting at 8 am on day 1, a hospital grade breast pump will be used to drain both breasts as confirmed by the absence of milk flow for 2 min during each episode of pumping and by palpation. Pumping will be performed in this manner every 3 hours around the clock. Subjects will be allowed a 5 hour window to sleep, however, as long as the total number of pumping episodes equals 8 in 24 hours.

During the first episode of pumping, a baseline prolactin level will be drawn immediately before the start of a pumping and repeated at 10 min intervals for 60 min, and then every 30 min for a total of 3 hours to document the peak prolactin level. An intravenous line will be placed to draw blood. Subsequently, subjects will be randomized to receive prolactin or placebo. On the morning of days 2, 5 and 8, blood will be collected for a prolactin level before medication injection. Subsequently, prolactin 60 mg/kg or placebo will be injected subcutaneously by the study nurse 3 hrs after the last pumping episode. On days 2 and 8, additional blood will be collected every 10 min for the first hour, every 30 min for hour 2 and 3, then at 4, 6 and 8 hours after injection to determine the peak prolactin level during a pumping session. Subjects will then drain both breasts as confirmed by the absence of milk flow for 2 min during each episode of pumping and by palpation and milk volume recorded. The subjects' vital signs will be monitored immediately before and every 15 minutes for 1 hr, every 30 min for hours 2 and 3, and then at 4, 6 and 8 hours after injection of prolactin/placebo. Temperature will be measured before the injection, every hour for hours 2 and 3, and then at 4, 6 and 8 hours after injection of placebo/prolactin. If there are no changes in vital signs, on days 5 and 8 vital signs will be monitored at baseline, only. Subjects will be taught to do SC injections on their own and will administer their second dose of SC r-hPRL or placebo 12 hours after the first dose. Subjects will continue every 12 hour SC r-hPRL or placebo administration for the next 7 days. Subjects will be asked to refrigerate all milk and bring it in to GCRC visits so that the volume that is recorded can be confirmed and for testing the milk composition and prolactin level before it is given to the infants. The final prolactin injection will be given on the evening of study day 8. All side effects in the mother and baby will be recorded daily throughout the study. Subjects will return for a final outpatient visit on day 16, to determine if any treatment effect persists. During this visit, milk will be pumped at baseline and volume recorded. In addition, blood will be drawn at 10 min intervals for 60 min, and then every 30 min for a total of 3 hours to document the peak prolactin level. Subjects will turn in their pumping diary the next day.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women, aged 18-45 years
* Lactation insufficiency postpartum
* Subjects will be women with children in the neonatal Intensive Care Unit (ICU) who are pumping breast milk for their infant's nutritional support and to maintain their milk supply.
* Subjects will have given birth at a gestational age of at least 24 weeks, and will generally be recruited 4-8 weeks postpartum.

Exclusion Criteria:

* Medications known to increase prolactin
* Anatomical breast abnormalities
* Use of medication contraindicated in breastfeeding mothers
* Allergies to mannitol
* Current use of hormonal contraception
* Previous mammoplasty or breast augmentation, unless they have successfully nursed an infant for 3 months in the past without requiring supplemental formula.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 11 (Actual)
Dates: Start 2004-09; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corrine K Welt, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Powe CE, Puopolo KM, Newburg DS, Lonnerdal B, Chen C, Allen M, Merewood A, Worden S, Welt CK. Effects of recombinant human prolactin on breast milk composition. Pediatrics. 2011 Feb;127(2):e359-66. doi: 10.1542/peds.2010-1627. Epub 2011 Jan 24. PMID 21262884

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2004-2008 Academic Hospital, clinical research center
Groups:
- Placebo Twice Per Day: Placebo group
  Normal Saline : twice per day
- Recombinant Human Prolactin Twice Per Day: Recombinant human prolactin every 12 hours
  Recombinant Human Prolactin : 60 mcg/kg every 12 hours
- Recombinant Human Prolactin Alternating With Placebo: Recombinant human prolactin alternating with placebo every 12 hours
  Recombinant human prolactin : 60 mcg/kg given every 24 hours alternating with normal saline placebo given once every 24 hours
Period: Overall Study
Arm/Group | Placebo Twice Per Day | Recombinant Human Prolactin Twice Per Day | Recombinant Human Prolactin Alternating With Placebo
Started | 4 | 4 | 3
Completed | 4 | 3 | 3
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: One subject did not complete the study and data was not analyzed for that subject.
Groups:
- Recombinant Human Prolactin Once Per Day: Recombinant human prolactin alternating with placebo every 12 hours
  Recombinant human prolactin : 60 mcg/kg given every 12 hours or every 24 hours
- Total: Total of all reporting groups
Arm/Group | Placebo Twice Per Day | Recombinant Human Prolactin Twice Per Day | Recombinant Human Prolactin Once Per Day | Total
Number analyzed (Participants) | 4 | 3 | 3 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 3 | 10
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (5) | 30 (5) | 32 (6) | 32 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 3 | 10
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Breast Milk Volume Baseline to 7 Days
Time Frame: 7 days
Measure: Mean (Standard Error); unit: % change from baseline
Groups:
- Recombinant Human Prolactin Alternating With Placebo: Recombinant human prolactin alternating with placebo every 12 hours
  Recombinant human prolactin : 60 mcg/kg given every 24 hours Placebo given every 24 hours
Arm/Group | Placebo Twice Per Day | Recombinant Human Prolactin Twice Per Day | Recombinant Human Prolactin Alternating With Placebo
Number analyzed (Participants) | 4 | 3 | 3
% change from baseline | -12 (27) | 429 (338) | 44 (28)

2. Secondary Outcome: Breast Milk Prolactin Levels
Time Frame: 7 days
Measure: Mean (Standard Error); unit: mcg/L
Arm/Group | Placebo Twice Per Day | Recombinant Human Prolactin Twice Per Day | Recombinant Human Prolactin Alternating With Placebo
Number analyzed (Participants) | 4 | 3 | 3
mcg/L | 60 (13) | 118 (25) | 118 (25)

ADVERSE EVENTS:
Arm/Group | Placebo Twice Per Day | Recombinant Human Prolactin Twice Per Day | Recombinant Human Prolactin Once Per Day
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/3
Other Adverse Events (participants affected / at risk) | 3/4 | 1/4 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Twice Per Day (N=4) | Recombinant Human Prolactin Twice Per Day (N=4) | Recombinant Human Prolactin Once Per Day (N=3)
Red marks (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Tiredness (General disorders) | 2 (2) | 1 (1) | 1 (1)
headache (General disorders) | 0 (0) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Menses (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes